CLINICAL TRIAL: NCT01571648
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Pharmacokinetics and Tolerability of Oral Azacitidine in Japanese Subjects With Myelodysplastic Syndromes
Brief Title: A Phase 1 Study to Evaluate the Pharmacokinetics and Tolerability of Oral Azacitidine in Japanese Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA-MDS-005
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral azacitidine (Experimental)
  Interventions: Drug: Oral azacitidine

INTERVENTIONS:
Drug: Oral azacitidine — Patients will receive 300 mg dose of oral azacitidine administered once daily for the first 21 days of each 28-day treatment cycle.

SUMMARY:
The purpose of this study is to evaluate the tolerability of oral azacitidine in the treatment of patients with Myelodysplastic Syndromes (MDS).

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following criteria to be enrolled in the study:

* Have a documented diagnosis of myelodysplastic syndromes (MDS) according to World Health Organization (WHO) 2008 classification
* Age ≥ 20 years;
* Written informed consent;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Resolution of any toxic effects of prior anti-cancer therapy; and
* Negative urine or serum pregnancy test on females of childbearing potential.

Exclusion Criteria:

The presence of any of the following will exclude a patient from enrollment:

* Treatment with chemotherapy, radiotherapy, or surgery within 4 weeks of study registration;
* Pregnant or breast-feeding females;
* Previous or concomitant malignancy other than MDS;
* Significant active cardiac disease within the previous 6 months;
* Uncontrolled systemic infection or
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity in accordance with Common Terminology Criteria for Adverse Events | 1 month
  Incidence of dose-limiting toxicity in accordance with Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
PK- Maximum concentration in plasma (Cmax) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK- Maximum concentration in plasma (Cmax)
PK- Time to maximum plasma concentration (Tmax) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK- Time to maximum plasma concentration (Tmax)
PK-Elimination rate constant (Kel) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK-Elimination rate constant (Kel)
PK-Terminal half-life (T1/2,z) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK-Terminal half-life (T1/2,z)
PK-Area under the plasma concentration-time curve (AUC) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK-Area under the plasma concentration-time curve (AUC)
PK-Apparent total body clearance (CL/F) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK-Apparent total body clearance (CL/F)
PK-Apparent volume of distribution (Vz/f) | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 hours post-dose
  PK-Apparent volume of distribution (Vz/f)
Safety (type, frequency, severity, number of participants with adverse events) | Up to 2 years
  Safety (type, frequency, severity, number of participants with adverse events)
Efficacy (Hematologic response and hematologic improvement) | Up to 2 years
  Efficacy (Hematologic response and hematologic improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Masamitsu Harata, Study Director — Celgene K.K.
Locations (5):
- Japan (5):
  - Celgene Trial Site, Fukuoka
  - Celgene Trial Site, Hiroshima
  - Celgene Trial Site, Nagoya
  - Celgene Trial Site, Osaka
  - Celgene Trial Site, Tokyo